CLINICAL TRIAL: NCT06407258
Title: Transdiagnostic Sleep Intervention Combined With Physical Activity Counseling (SLEEPAC) in Adolescent Psychiatric Patients: A Blended Care Approach
Brief Title: Promoting Sleep and Physical Activity Among Adolescent Psychiatric Patients
Acronym: SLEEPAC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christin Lang (Other)
Collaborators: Department of Sport, Exercise, and Health, University of Basel (Unknown); University Hospital of Child and Adolescent Psychiatry and Psychotherapy (Unknown); University Children's Hospital of Basel (Unknown); Psychiatry Baselland (Unknown)
Responsible Party: Sponsor-Investigator, Christin Lang, PhD, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLEEPAC
Record Dates: First submitted 2024-04-30; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Mental Disorder in Adolescence; Insomnia; Delayed Sleep-Wake Phase Disorder
Keywords: adolescents; CBT-I; light therapy; circadian adaptation; physical activity counseling; transdiagnostic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SLEEPAC (Experimental): In addition to treatment-as-usual (TAU), participants of the SLEEPAC arm will receive a multi-component sleep intervention combining elements of CBT-i, circadian adaptation, and physical activity counselling.
  Interventions: Behavioral: SLEEPAC
- Control (No Intervention): Participants of the control group continue with their treatment as usual

INTERVENTIONS:
Behavioral: SLEEPAC — 6x individual blended-care counselling sessions:
  * 1 x face-to-face kick-off sessions at study site (45 min)
  * 1 x try-out exercise sessions at study site (45 min)
  * 4 x online face-to-face sessions via zoom (30 min)
  * Both the intervention and the waitlist control condition will continue with TAU.
  Component 1: CBT-I: Sleep restriction, and cognitive therapy strategies with education about sleep-wake regulation, sleep hygiene, and pre-bedtime counter arousal methods.
  Component 2: Circadian treatment: Morning bright light therapy with a gradual advanced sleep schedule and timed morning exercise.
  Component 3: Physical activity counselling involves providing personalized guidance and support to individuals to help them adopt and maintain a physically active lifestyle tailored to their preferences and needs.
  Arms: SLEEPAC

SUMMARY:
Mental health disorders pose a significant burden on adolescent populations globally, often accompanied by sleep disturbances. Emerging evidence suggests that addressing sleep issues can improve mental health outcomes, while physical activity is increasingly recognized as beneficial for both sleep and mental well-being. This study aims to assess the effectiveness of a novel intervention (SLEEPAC), combining cognitive-behavioral therapy for insomnia (CBT-I), circadian treatment, and PA counseling, compared to treatment as usual (TAU), in improving psychopathology among adolescent psychiatric outpatients with sleep disturbances. Secondary outcomes include improvements in sleep health, physical activity levels, cognitive performance and self-esteem. Additionally, the study seeks to explore the predictive value of sleep neurophysiological biomarkers using high-density sleep electroencephalography (EEG), contributing to advancements in precision psychiatry for this population.

DETAILED DESCRIPTION:
Background and rationale. Mental health disorders are the leading cause of disability in adolescents worldwide. 70 to 80% of individuals with mental disorders experience sleep disturbances. Preliminary evidence from adult studies suggest that treating sleep disturbances in these patients can improve mental health outcomes. Moreover, regular physical activity (PA) is increasingly promoted as a remedy for sleep and other mental health problems. Thus, combining sleep therapy and PA counseling may synergistically improve mental health outcomes in adolescent psychiatric patients. Guidance on how to address sleep disturbances and PA counselling among this population in routine clinical care has the potential to improve clinical and psychosocial outcomes.

Overall objectives. To improve psychopathology in adolescent psychiatric outpatients with comorbid sleep disturbances by testing a novel behavioral intervention (TRANSPAC) that improves both sleep and PA levels. This multi-component intervention combines CBT-I, circadian treatment, and PA counseling and will be compared against treatment as usual (TAU).

Specific aims. With the prospect of further developing and fine-tuning transdiagnostic treatment protocols for young psychiatric patients with comorbid sleep disturbances, the objectives of the proposed study are twofold: (1) To test the efficacy of a novel transdiagnostic blended care e-health sleep (CBT-I + circadian treatment) and PA therapy and to test its efficacy against TAU. The primary endpoint is severity reduction of psychopathology. Improvements of sleep health and regular PA levels will be investigated as secondary outcomes. (2) To evaluate the prognostic value of sleep neurophysiological biomarkers (high-density sleep-EEG) on intervention efficiency, thereby advancing current approaches in precision psychiatry.

Methods. The proposed study will recruit 140 psychiatric outpatients with comorbid sleep problems from our partner clinics in Basel and Bern (KJP-UPD Bern, UKBB Basel). Inclusion criteria: aged 13-18 years, presence of sleep problems in addition to a psychiatric diagnosis. Adolescents will be serially randomized over 1,5 years into one of 2 intervention arms: (a) TRANSPAC; or (b) TAU. The intervention will be delivered in 6 sessions over 12 weeks. Data will be collected at 3 time points: Baseline, post-intervention, and 6-months follow-up. Psychopathological load will be assessed via Symptom Checklist-90-Revised. The composite sleep health score is based on self-reported sleep quality, -quantity, and timing, complemented by 7-day sleep tracker (Oura Ring Gen3). PA will be assessed objectively via the same device (Oura Ring was selected due to prior compliance issues among this population with Actigraph). Primary biomarkers are the micro-architectural features of sleep assessed by a high-density sleep-EEG, such as sleep spindles, slow wave activity, and REM-latency. Secondary biomarkers include heart rate variability, and fitness.

Expected results. The proposed study aims to further develop and fine-tune transdiagnostic treatment protocols (i.e. for multiple psychiatric disorders) in adolescent psychiatric outpatients with sleep disturbances. Testing the potential of sleep treatments for improving psychopathology in young psychiatric patients is a promising and highly novel approach. Thus, it is expected that both TRANSPAC and TAU will improve psychopathology in youth, with TRANSPAC resulting in superior effects than TAU alone.

Impact. The onset of mental health disorders is often during adolescence, requiring countermeasures at an early developmental stage. Since sleep disturbances are a diagnostic feature for many psychiatric disorders, treating sleep problems transdiagnostically may positively impact other health outcomes. PA counseling may complement the benefits of the sleep intervention, working in concert to improve mental health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 13 to 18 years
* Presence of insomnia and/or delayed sleep-wake phase disorder
* At least one further diagnosis of DSM-5
* Written informed consent of parents / primary caregiver

Exclusion Criteria:

* Organic sleep- and brain disorders (i.e., obstructive sleep apnea, narcolepsy, epilepsy)
* Suffering from medical conditions, which prevent participation in physical activity
* Changes to medication regime during the study protocol
* Color-blindness (due to stroop test)

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Psychopathology | 10 minutes
  Symptom Checklist-90-Revised (SCL-90-R) is one of the most comprehensive and widely used questionnaires to assess psychopathology. It is validated for youth psychiatric inpatients from age 13 onwards. The Symptom Checklist contains a list of problems and complaints that people sometimes have. Participants are asked how much they were bothered by that problem during the past week. Answers range from 0=not at all to 4=extremely. Thus, a higher factor score indicated more serious psychiatric symptoms problems.

SECONDARY OUTCOMES:
Composite Sleep Health | 10-20 min (questionnaire), 7 days (sleep tracker Oura Gen3)
  The use of a single disorder-focused sleep measure might be problematic to capture intervention effects among a transdiagnostic sample. A composite sleep health score comprising 6 dimensions of sleep and circadian functioning (daytime alertness, sleep satisfaction, -timing, -efficiency, -duration, and -regularity) was found to predicted mental health in adolescents. Using these components, a weighted summary sleep health score will be calculated, based on results from exploratory factor analyses.
  The following questionnaires will be used:
  The Pittsburgh Sleep Quality Index (PSQI) The Pediatric Daytime Sleepiness Scale (PDSS) The Sleep condition indicator (SCI) 7-day Habitual sleep-wake pattern (Oura Ring Gen3) Children's Morningness-Eveningness Preference Scale (CMEP) Munich Chronotype Questionnaire (MCTQ)
  According to LuDong et al. 2019, each dimension will be dichotomized as "good" (=1) or "poor" (=0). Thus a higher score indicates better sleep health.
Physical Activity | 7 days
  Habitual physical activity patterns will be captured with the Oura Ring Gen3. For 7 consecutive days and nights, participants will wear the small finger ring on their non-dominant hand over 7 days and nights to collect objective physical activity patterns. Additionally, a 7-day physical activity recall will be conducted at the end of the week with a trained staff member.
Cognitive performance | 10 min
  Cognitive Performance will be assessed with a modified version of the Stroop task, which includes trials demanding inhibitory control and emotion recognition. The computer-based task is administered with E-Prime 3.0 (PST, USA). Participants complete testing in a seated position, with a viewing distance of approximately 80 cm. Assessments are performed in a dimly lit room at an environmental temperature of 21-22 °C. The surrounding noise is reduced to a minimum and participants are instructed to avoid movements and noise during cognitive testing. The testing sequence is identical for all participants and lasts 10 to 15 min.
Self-esteem | 5 min
  Self-esteem will be assessed with the Rosenberg Self-Esteem Scale

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Department of Sport, Exercise, and Health, University of Basel, Basel, Canton of Basel-City
  - University Hospital of Child and Adolescent Psychiatry and Psychotherapy, Bern, Canton of Bern

IPD SHARING:
Plan to Share IPD: No